CLINICAL TRIAL: NCT02769624
Title: A Randomized, Placebo-Controlled Pilot Study to Determine the Acute Effects of Inhaled Treprostinil on Exercise, Vascular Function, and Exercise Induced Liver Stiffness in Fontan Patients
Brief Title: Acute Effects of Inhaled Treprostinil in Fontan Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped early due to inability to recruit additional participants
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2015-1491
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treprostinil (Experimental): A dose of 18mcg (3 breaths) will be administered using the Tyvaso® (treprostinil) inhalation system. Tyvaso® (treprostinil) inhalation solution is supplied in 2.9 mL clear ampules packaged as four ampules in a foil pouch. Frequency and duration- 3 times over 1 study visit.
  Interventions: Drug: Treprostinil
- Placebo (Placebo Comparator): A dose of 3 breaths of placebo will be administered using the Tyvaso® (treprostinil) inhalation system. Placebo will be supplies in matching ampules to treprostinil. Volume will match that of treprostinil. Frequency and duration- 3 times over 1 study visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil — A dose of 18mcg (3 breaths) will be administered 3 times: at baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
  Other Names: Tyvaso
  Arms: Treprostinil
Drug: Placebo — 3 breaths of placebo (via inhalation devices) will be administered 3 times: at baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
  Arms: Placebo

SUMMARY:
In this pilot study investigators propose to explore the effects of a locally delivered inhaled pulmonary vasodilator (inhaled treprostinil) on exercise performance, pulmonary blood flow, venous pressure response and vascular function in stable Fontan patients. Investigators will also assess the effects of resting and acute rises in exercise induced systemic venous pressure on liver stiffness and will also assess whether treprostinil will attenuate the acute stiffness increase that investigators expect to see. This will be a prospective, randomized, double-blinded placebo controlled, crossover trial. Following recruitment and informed consent, each participant will undergo three study visits, including baseline testing (visit 1), followed by two sets of exercise and vascular function tests (visit 2 and visit 3) at CCHMC. Twenty-six patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years and older
2. Single ventricle patients status post Fontan procedure

Exclusion Criteria:

1. Clinically unstable: these are patients who are experiencing new cardiovascular symptoms such as worsening shortness of breath, new onset arrhythmia, uncontrolled heart failure, or evidence of clinically significant cirrhosis or renal failure.
2. Evidence of Fontan pathway or intra cardiac obstruction as identified on prior clinically indicated imaging studies (echocardiography and MRI);
3. Evidence of left or right systemic ventricular systolic dysfunction with an Ejection fraction of <40% on either echocardiogram or MRI from previously documented clinical data;
4. Presence of uncontrolled arrhythmias;
5. Unable to perform exercise testing for any reason or if deemed by the PI or designee that exercise testing would not be in the best interest of the participant
6. Currently pregnant and/or breastfeeding
7. Patient unable to provide informed consent
8. BMI > 30 mg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gruschen Veldtman, MBChB, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, double-blind, crossover trial conducted at one center. Healthy Fontan patients were recruited from within the medical center's Fontan management program for participation in this trial. Each patient completed three study visits over the course of six weeks.
Pre-assignment Details: Each participant came in for a baseline visit initially and then for the second visit, they were randomly assigned to receiving either the study medication or placebo. At the third visit, the patient received the opposite of what they received at visit two.
Groups:
- Treprostinil, Then Placebo; Placebo, Then Treprostinil: A dose of 18mcg (3 breaths) will be administered using the Tyvaso® (treprostinil) inhalation system. Tyvaso® (treprostinil) inhalation solution is supplied in 2.9 mL clear ampules packaged as four ampules in a foil pouch. Frequency and duration- 3 times over 1 study visit.
  Treprostinil: A dose of 18mcg (3 breaths) will be administered 3 times: at baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
  A dose of 3 breaths of placebo will be administered using the Tyvaso® (treprostinil) inhalation system. Placebo will be supplies in matching ampules to treprostinil. Volume will match that of treprostinil. Frequency and duration- 3 times over 1 study visit.
  Placebo: 3 breaths of placebo (via inhalation devices) will be administered 3 times: at baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
Period: Overall Study
Arm/Group | Treprostinil, Then Placebo | Placebo, Then Treprostinil
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Fifteen participants began the study, however, only 14 completed both the study medication and placebo components of the trial.
Groups:
- Treprostinil Crossover With Placebo: Participants may receive either treprostinil or placebo at visit 2. They will receive the opposite at visit 3.
  If receiving treprostinil, a 18mcg dose (3 breaths) will be administered using the Tyvaso® (treprostinil) inhalation system. Tyvaso® (treprostinil) is supplied in 2.9 mL clear ampules packaged as four ampules in a foil pouch. Frequency and duration- 3 times over 1 study visit: baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
  If receiving placebo, a dose of 3 breaths of placebo will be administered using the Tyvaso® (treprostinil) inhalation system. Placebo will be supplied in matching ampules to treprostinil. Volume will match that of treprostinil. Frequency and duration- 3 times over 1 study visit: baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
Arm/Group | Treprostinil Crossover With Placebo
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14
Cardiac Anatomy [Count of Participants; unit: Participants]
  Tricuspid Atresia | 4
  Double Inlet Left Ventricle | 2
  Pulmonary Atresia | 2
  Hypoplastic Left Heart Syndrome | 6
Fontan Type [Count of Participants; unit: Participants]
  Atrio-pulmonary Fontan | 2
  Lateral Tunnel | 9
  Extracardiac Conduit | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Liver Stiffness Through the Measurement of Shear Wave Ultrasound Elastography (m/s)
Description: At rest and then following maximal exercise, shear wave ultrasound elastography will be performed to assess if the study medication shows an improvement in liver stiffness (reduction in m/s number) following maximal exercise versus at rest.
Time Frame: At rest and following dose 2
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
m/s
  Rest | 2.39 (0.67) | 2.38 (0.71)
  Following maximal exercise | 2.79 (0.54) | 2.89 (0.51)

2. Secondary Outcome: Venous Pressure (mmHg) at Rest and Peak Exercise
Description: Venous pressure was measured both at rest and during an incremental ramp exercise test. Comparison was made to evaluate if the treprostinil study medication had a different effect in venous pressure measurements during peak exercise versus placebo.
Time Frame: At rest and at peak incremental exercise
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
mmHg
  Rest | 12.8 (3.08) | 12.1 (2.43)
  Peak Incremental Exercise | 22.8 (6.16) | 22.6 (8.04)

3. Secondary Outcome: Exercise Endurance Time (in Minutes)
Description: A constant work rate exercise test will be performed to determine exercise endurance
Time Frame: Immediately following dose 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
Minutes | 5.19 (0.89) | 5.82 (1.23)

4. Secondary Outcome: Peak Volume of Oxygen Consumption (VO2) (ml/kg/Min)
Description: Measuring the difference in peak/maximal VO2 during incremental exercise testing to assess if the response during peak exercise is different when utilizing treprostinil versus a placebo.
Time Frame: Maximal exercise test (5-10 minutes)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
ml/kg/min | 23.4 (6.67) | 24.6 (9.04)

5. Secondary Outcome: Minute Volume and Carbon Dioxide Volume Slope (VE/VCO2) During Incremental Exercise
Description: Measuring the difference in peak/maximal VE/VCO2 during incremental exercise testing to assess if the response during peak exercise is different when utilizing treprostinil versus a placebo. The VE/VCO2 slope is used to show the relationship between minute ventilation and carbon dioxide production.
Time Frame: Maximal exercise test (5-10 minutes)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
unitless | 26.8 (4.95) | 26.1 (6.35)

6. Secondary Outcome: VO2 (ml/kg/Min) at Anaerobic Threshold
Description: Measuring the difference in VO2 at anaerobic threshold of an incremental exercise test to assess the variance in response with treprostinil versus placebo
Time Frame: Maximal exercise test (5-10 minutes)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Treprostinil | Placebo
Number analyzed (Participants) | 14 | 14
ml/kg/min | 17.3 (3.63) | 18.1 (5.36)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed and recorded following signing of informed consent through two weeks following the last study visit (period ranging from 6-9 weeks).
Description: Events that are unexpected and considered to be related or possibly related to the study procedures as well as breaches of confidentiality, and protocol violations were reported to the IRB as soon as possible after discovery of the event. All adverse events will be classified by the PI for relationship, severity, and expectedness. Events not meeting the criteria for prompt reporting were reported to the Institutional Review Board (IRB) at the time of continuing review.
Groups:
- Treprostinil; Placebo: Participants may receive either treprostinil or placebo at visit 2. They will receive the opposite at visit 3.
  If receiving treprostinil, a 18mcg dose (3 breaths) will be administered using the Tyvaso® (treprostinil) inhalation system. Tyvaso® (treprostinil) is supplied in 2.9 mL clear ampules packaged as four ampules in a foil pouch. Frequency and duration- 3 times over 1 study visit: baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
  If receiving placebo, a dose of 3 breaths of placebo will be administered using the Tyvaso® (treprostinil) inhalation system. Placebo will be supplied in matching ampules to treprostinil. Volume will match that of treprostinil. Frequency and duration- 3 times over 1 study visit: baseline, 1.5 hrs. post baseline and then again 2 hrs later following maximal exercise testing.
Arm/Group | Treprostinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 11/14 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil (N=14) | Placebo (N=15)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 0 (0)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Increase in Liver Lab Values (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abnormal ECG Rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Weakness (General disorders) | 1 (1) | 1 (1)
Lowered blood pressure (Cardiac disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study had a small sample size and may have had selection bias towards well-functioning Fontan patients, who might benefit less from the use of pulmonary vasodilators. Additional physiological factors could have been assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT02769624/Prot_SAP_000.pdf